CLINICAL TRIAL: NCT05343013
Title: TAS-102 With or Without Celecoxib in ctDNA-defined Minimal Residual Disease in Colorectal Cancer After Completion of Adjuvant Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Taiho (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0823; NCI-2022-03438 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-04-15; First posted 2022-04-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Trifluridine; tipiracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS-102 (Experimental): TAS-102 should be taken by mouth 2 times a day, within 1 hour after your morning and evening meals (about 12 hours apart).
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102 — GIven by PO
  Other Names: trifluridine; tipiracil; Lonsurf

SUMMARY:
To measure the level of circulating tumor DNA (ctDNA) in the blood of colorectal cancer patients after 6 months of receiving TAS-102 therapy. ctDNA is genetic material from tumor cells that can be found and measured in the blood.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective is to determine the 6-month ctDNA clearance rate in colorectal cancer patients with minimal residual disease following 6 months of TAS-102 therapy.

Secondary Objectives:

* To determine the 3-month ctDNA clearance rate in colorectal cancer patients with minimal residual disease.
* To determine the disease free survival (DFS) amongst colorectal cancer patients with minimal residual disease following 6 months of TAS-102 therapy.
* To determine the overall survival (OS) amongst colorectal cancer patients with minimal residual disease following 6 months of TAS-102 therapy.
* To determine the safety and tolerability of TAS-102 for the treatment of colorectal cancer patients with minimal residual disease.

Exploratory Objectives:

* To determine markers of response and resistance in archival tumor tissue including but not limited to immune profiles of tumor-infiltrating lymphocytes, expression of immune markers in tumor cells and microenvironment, and molecular markers (including but not limited to mutations, deletions, and/or amplifications or cancer molecular subtype)
* To determine changes in profiles of circulating lymphocytes and ctDNA with treatment
* To determine baseline characteristics in archival tumor and/or plasma that may predict clinical benefit

ELIGIBILITY:
Inclusion Criteria:

1. Has histological confirmation of colorectal cancer
2. Received post-R0 resection of stages II, III, or IV colorectal cancer and has completed all planned curative intent therapies that must include ≥ 3 months of oxaliplatin containing chemotherapy
3. Has no definitive evidence of radiographic disease per assessment by investigators within 28 days (before or after) a positive ctDNA assay
4. Has minimal residual disease as defined by positive ctDNA assay (completed as standard-of-care at MD Anderson). Patients may be identified for enrollment with any Clinical Laboratory Improvement Amendments (CLIA)-certified ctDNA assay for MRD. MRD status will be confirmed with the Signatera assay prior to initiation of therapy (unless the prior testing was also done with Signatera in which case this test would not require confirmation)
5. Has adequate organ and marrow function as defined below:

   1. absolute neutrophil count: ≥1,000/mcL
   2. platelets: ≥100,000/mcL
   3. total bilirubin: ≤ institutional upper limit of normal (ULN)
   4. AST(SGOT)/ALT(SGPT): ≤3 × institutional ULN
   5. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥60 mL/min. Creatinine clearance (Clcr) can either be measured in a 24-hour urine collection or estimated by the Cockcroft-Gault equation as follows: Clcr (mL/min) = [(140 - age) x (weight in kg) ÷ [72 x (serum creatinine in mg/dL)] [0.85 if female]
6. Has ECOG performance status (PS) of 0 or 1
7. Is of age ≥ 18 years. Because no dosing or adverse-event data are currently available on the use of TAS-102 in patients, children <18 years of age are excluded from this study.
8. Is able to understand and is willing to sign a written informed consent document.
9. Is willing to utilize contraception. Female subjects agree to use highly effective contraception combined with an additional barrier method (eg, diaphragm, with a spermicide) while on study and for 7 months after last dose of study drug, and the same criteria are applicable to male subjects if they have a partner of childbirth potential. Male subject agrees to use a condom and not donate sperm while in this study and for 7 months after the last treatment.

Exclusion Criteria:

1. Has other concomitant active, invasive malignancies that may interfere with ctDNA analysis (known clonal hematopoesis of unknown potential allowed)
2. Has serum electrolytes, potassium, calcium, or magnesium levels outside of the normal laboratory reference range which are clinically significant in the investigator's judgment
3. Has significant concomitant health conditions including but not limited to severe autoimmune or cardiovascular disorders that may interfere with participation in the study per assessment by investigators
4. Has a persistent adverse event, except alopecia and neuropathy, greater than or equal to grade 2 of the Common Toxicity Criteria for Adverse Events (CTCAE) v. 5.0
5. Has another disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition that investigators suspect may (a) prohibit use of the investigational product, (b) affect interpretation of study results, or (c) put the patient at undue risk of harm
6. Has known hypersensitivity to the trial drugs or their excipients or is at risk of allergic of anaphylactic reaction to drug product according to the Investigator's judgement
7. Is pregnant or lactating
8. Is unable to take medication orally or has any other condition that investigators believe may affect absorption of the investigational product
9. Is receiving any other investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
To determine the 6-month ctDNA clearance rate in colorectal cancer patients with minimal residual disease following 6 months of TAS-102 therapy. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alisha Bent, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pellatt AJ, Bent A, Hornstein N, Parseghian C, Huey R, Raghav K, Morris V, Overman M, Morelli P, Willis J, Le P, Shen JP, Kee B, Eluri M, Higbie V, Alfaro-Munoz K, Aziz K, Kell R, Sun R, Kopetz S, Dasari A. Phase II Trial of TAS-102 in Colorectal Cancer Patients With Circulating Tumor DNA-Defined Minimal Residual Disease After Adjuvant Therapy: INTERCEPT-TT. JCO Precis Oncol. 2025 Jul;9:e2500142. doi: 10.1200/PO-25-00142. Epub 2025 Jul 16. PMID 40669021
- See also: M D Anderson Cancer Center — http://www.mdanderson.org